CLINICAL TRIAL: NCT07150871
Title: Impact of the COVID-19 Pandemic on Syphilis: Epidemiological Changes and Interaction With HIV
Brief Title: Impact of Covid-19 on Syphilis
Acronym: SIPAND
Status: Active, not recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.Minf.25.01
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Syphilis; COVID - 19; HIV (Human Immunodeficiency Virus); Retrospective Studies
MeSH Terms: conditions — Syphilis; COVID-19; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients diagnosed with syphilis — Collection of clinical data from patients aged ≥18 years with a microbiological and/or clinical diagnosis of syphilis, treated by the Infectious Diseases Department of the University Hospital of Alessandria from 2017 to 2025.

SUMMARY:
Sexually transmitted infections (STIs) represent a significant challenge to global public health. Although many of these infections are treatable, failure to diagnose and delayed treatment can lead to serious complications, including infertility, chronic inflammatory diseases, and an increased risk of HIV transmission. The COVID-19 pandemic has had a significant impact on healthcare management, the economy, and citizens' lifestyles. The first lockdown in the spring of 2020 affected the entire country, while in the following months, government measures were differentiated on a regional basis, with varying restrictions on activities and mobility. Physical distancing, the use of personal protective equipment, fear of contagion, and health restrictions contributed to a delay in STI diagnoses, resulting in an increase in transmission and severity of cases diagnosed after 2022.

DETAILED DESCRIPTION:
Syphilis is a chronic infectious disease with a prolonged course, characterized by considerable clinical variability, so much so that it is referred to as the great imitator, due to its ability to manifest itself with symptoms that can mimic numerous other diseases. The clinical picture develops through alternating phases of activity, with obvious symptomatic manifestations, and latency, in which the infection remains silent in the body. It is a globally widespread infection, transmitted mainly through sexual contact, although it can also be transmitted congenitally or through direct contact with infected lesions. The relationship between syphilis and HIV is of growing clinical importance due to increasing rates of co-infection and the particular interaction between these two STIs. Syphilis facilitates the transmission and acquisition of HIV, while HIV infection accelerates the natural progression of syphilis. In addition, HIV has been associated with false positive and false negative results in serological tests for syphilis, complicating the diagnosis and management of the disease. A study conducted by the Department of Medicine in Toronto and the Ministry of Health showed that, in individuals with latent syphilis, the prevalence of HIV remained stable between 1991 and 2012, but increased approximately fivefold from 2012 to 2020, reaching a peak of 52.6%. In 2022, the Ministry of Health reported that syphilis cases had doubled compared to 2018, with incidence rising from 2.5 to 4.3 cases per 100,000 inhabitants. Gonorrhea increased from 1.5 to 3.3 cases per 100,000 inhabitants during the same period. Chlamydia, although less documented than in other European countries, also showed an upward trend, with 1,396 cases per 100,000 inhabitants in 2022. The COVID-19 pandemic has had a significant impact on healthcare management, the economy, and citizens' lifestyles. The first lockdown in the spring of 2020 affected the entire country, while in the following months, government measures were differentiated on a regional basis, with varying restrictions on activities and mobility. Physical distancing, the use of personal protective equipment, fear of contagion, and health restrictions contributed to a delay in STI diagnoses, resulting in an increase in transmission and severity of cases diagnosed after 2022. A study published in BMJ Open in 2021 analyzed the impact of the pandemic on healthcare services compared to previous years. The systematic review highlighted a 37% reduction in access to care, with decreases of 42% for outpatient visits, 28% for hospitalizations, 31% for diagnostics, and 30% for therapies. The pandemic has therefore significantly reduced the use of healthcare services, with a greater impact on people with non-serious conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with microbiological and/or clinical diagnosis of syphilis
* Patients treated by the Infectious Diseases Department of the University Hospital of Alessandria
* Signature of informed consent form

Exclusion Criteria:

* Patients for whom the data required for the study are not available in medical records or electronic filing systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥18 years with a microbiological and/or clinical diagnosis of syphilis, treated by the Infectious Diseases Department of the University Hospital of Alessandria from 2017 to 2025
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Trend of syphilis | Baseline
  Analyze the trend of syphilis before and after the COVID-19 pandemic

SECONDARY OUTCOMES:
Characteristics of affected patients | Baseline
  Describe the characteristics of patients with syphilis referred to the Infectious Diseases Unit of the SS Antonio e Biagio e Cesare Arrigo University Hospital in Alessandria between 2017 and 2025.
Interaction between syphilis and HIV | Baseline
  Examine the interaction between syphilis and HIV in a post-pandemic context, identifying how the pandemic has affected co-infection between syphilis and HIV, monitoring any changes in co-infection rates.
Infection Recurrence Rate | Baseline
  Evaluate the infection recurrence rate, calculated by taking the date of recovery from the original infection as the baseline and the onset of the same infection as the event of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No